CLINICAL TRIAL: NCT06985576
Title: A Long-term Follow-up Study of GF-01-01 to Evaluate the Safety and Persistence of GF-CART01 (CD20/19 CAR T Cell) in Subjects With Relapsed or Refractory B-Cell Hematological Malignancies
Brief Title: Long-term Study to Evaluate Safety and Persistence of GF-CART01
Status: Not yet recruiting | Type: Observational
Sponsor: GenomeFrontier Therapeutics TW Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: GF-01-01e
Record Dates: First submitted 2025-05-15; First posted 2025-05-22 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: DLBCL - Diffuse Large B Cell Lymphoma; Follicular Lymphoma (FL); Primary Mediastinal Large B-Cell Lymphoma; High Grade B Cell Lymphoma
MeSH Terms: conditions — Dendritic Cell Sarcoma, Interdigitating; Lymphoma, Follicular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- LTFU: Subjects who participated in the initial study of GF-01-01 and received treatment with GF-CART01, irrespective of their completion status, are invited to participate in this follow-up study.

SUMMARY:
The goal of this observational study is to learn about the long-term safety of GF-CART01 after cell infusion up to 15 years.

DETAILED DESCRIPTION:
This comprehensive long-term follow-up study is meticulously designed to assess the safety and persistence of GF-CART01. Subjects who participated in the initial study of GF-01-01 and received treatment with GF-CART01, irrespective of their completion status, are eligible to participate in this follow-up study. The study may allow for a maximum enrollment of 18 subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects previously enrolled in the study of GF-CART01 (Protocol No.: GF-01-01) and received GF-CART01 infusion
2. Subjects or their legal guardians must volunteer to participate in the study and sign the informed consent
3. Willingness and ability to comply with protocol-stated requirements, instructions, and restrictions in the investigator's judgement

Exclusion Criteria: None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects who participated in the initial study of GF-01-01 and received treatment with GF-CART01, irrespective of their completion status, are eligible to participate in this follow-up study. The study may allow for a maximum enrollment of 18 subjects.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Estimated)
Dates: Start 2026-05 (Estimated); Primary Completion 2041-05 (Estimated); Study Completion 2041-05 (Estimated)

PRIMARY OUTCOMES:
Long-Term Safety of GF-CART01 after infusion | up to 15 years after GF-CART01 infusion
  Percentage of subjects with ≥ grade 3 GF-CART01-related adverse events, serious adverse events (SAEs), adverse events of special interest (AESIs)

SECONDARY OUTCOMES:
GF-CART01 persistence | up to 15 years after GF-CART01 infusion
  Measure the duration of GF-CART01 presence after cell infusion
  * Clast
  * Time of Clast
Efficacy of GF-CART01 | up to 15 years after GF-CART01 infusion
  Assess the overall survival (OS) up to 15 years after GF-CART01 infusion

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No